CLINICAL TRIAL: NCT05926063
Title: Stopping Antibiotics After 3 Days for the Treatment of FEbrile Neutropenia in Haematology Patients (SAFE Study): a Randomized Open-label Non-inferiority Trial
Brief Title: Stopping Antibiotics After 3 Days for the Treatment of High-risk FEbrile Neutropenia
Acronym: SAFE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Antwerp (Other); AZ Sint-Jan AV (Other); Centre Hospitalier Universitaire de Liege (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S66527; 2022-500389-84 (EudraCT Number)
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-06

CONDITIONS: Neutropenia, Febrile
Keywords: Neutropenia; Leukemia; Stem Cell Transplant Complications; Infections
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia; Leukemia; Infections

STUDY DESIGN:
Intervention Model Description: Comparison of two treatment strategies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short treatment group (Experimental): Empirical broad-spectrum antibiotics (EBAT) as per local protocol:
  * Meropenem 3 x 1(/2) g IV; OR
  * Piperacilline-Tazobactam 4 x 4 g IV; OR
  * Cefepime 3 x 2 g IV; OR
  * Ceftazidim 3 x 2 g IV
  Short treatment group: EBAT will be discontinued:
  * After 3x24 hours;
  * Irrespective of presence of fever; AND
  * If no clinical of microbiological infection is documented.
  Interventions: Other: Comparison short vs extended EBAT treatment group
- Extended treatment group (Active Comparator): Empirical broad-spectrum antibiotics (EBAT) as per local protocol:
  * Meropenem 3 x 1(/2) g IV; OR
  * Piperacilline-Tazobactam 4 x 4 g IV; OR
  * Cefepime 3 x 2 g IV; OR
  * Ceftazidim 3 x 2 g IV
  Extended treatment arm: EBAT will be continued:
  * At least 5x24 hours;
  * Until afebrile (TMT<38.0°C) for at least 5 consecutive days; OR
  * Until resolution of neutropenia (ANC >0,5 x109/L); OR
  * Until they have been treated 10 days, whatever comes first.
  Interventions: Other: Comparison short vs extended EBAT treatment group

INTERVENTIONS:
Other: Comparison short vs extended EBAT treatment group — This study compares two management strategies of patients undergoing treatment with chemotherapy or a stem cell transplantation. One strategy is to treat these patients at the time of febrile neutropenia with a fixed 72 hours course of EBAT. The other, more commonly followed strategy is a longer minimum EBAT duration of 5 days as well as other variables like neutrophil recovery and defervescence. In both arms, definitive treatment is given when an infectious cause of the fever is found according to local guidelines (e.g. pneumonia or mucosits with bacteremia).

SUMMARY:
The goal of this clinical trial is to compare a short course of antibiotics in patients in whom no bacterial infection is found with the current "golden standard": long-term antibiotic treatment in adult hematology patients who develop neutropenic fever.

The main question it aims to answer is: whether the short-term treatment is equally safe for patients, hence the name 'SAFE study'.

Participants will be randomly assigned (randomized) to one of two treatment options once they develop neutropenic fever: short-term or long-term antibiotic treatment. An additional blood sample, urine sample and stool sample will be collected.

Researchers will compare the short-term and the long-term antibiotic treatment groups to see if the short treatment is equally safe as the long-term treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures;
* Age older than 16 years;
* Intensive therapy is started within three days before randomization for one of the following haematological conditions:

  * Remission induction chemotherapy for newly diagnosed acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS); OR
  * Re-induction chemotherapy for relapsed after haematological remission lasting for a minimum duration of 6 months; OR
  * Conditioning regimen to prepare for an allogeneic HCT; OR
  * Conditioning regimen to prepare for an autologous HCT.
* Expected longstanding (≥ 7 days) neutropenia (ANC < 0.5x10^9/L);
* Expected length of hospital stay of at least 10 days.

Exclusion Criteria:

1. Clinically or microbiologically documented infection;
2. Patient already receives broad spectrum antibiotic therapy;
3. Any critical illness for which Intensive Care Unit treatment is required;
4. SOFA score ≥ 11;
5. Longstanding neutropenia (>21 days) prior inclusion;
6. Previous enrolment in this study;
7. Not able to provide written informed consent;
8. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol;
9. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Absence of a serious medical complication (SMC) following 42 days after randomisation. SMC is defined as: Death; and/or ICU admission; and/or Septic shock requiring vasopressive therapy. | 42 days

SECONDARY OUTCOMES:
Incidence of bacteraemia within 42 days after randomisation | 42 days
Clinically documented infections | 42 days
Number of documented bacterial infections | 42 days
Total days of non-prophylactic antibiotics given to the patient at engraftment | 42 days
Total numbers of antibiotic switches before neutrophil recovery | 42 days
Incidence of Clostridium difficile infection | 42 days
Incidence, severity and duration of diarrhea | 42 days
Incidence of candidemia | 42 days
Length of hospital stay in the first 42 days after randomization | 42 days
Number of patients admitted to the ICU within 42 days after randomisation | 42 days
Number of readmissions within 42 days | 42 days
Number of patients with a culture (surveillance or diagnostic culture) positive for resistant bacteria: VRE; ESBL; MRSA; and/or CPE | 42 days
Duration of hospitalization | 42 days
Number of patients in the short treatment arm with ongoing fever at time of EBAT stop | 42 days
Incidence of acute GVHD (grade II or higher) in the transplanted study population | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Johan Maertens, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium